CLINICAL TRIAL: NCT01149941
Title: Randomized, 2-way Crossover, Bioequivalence Study of Ibuprofen 200 mg Gel Capsules and Advil Liquigels 200 mg Gel Capsules Administered as 1 x 200 mg Gel Capsules in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Ibuprofen 200 mg Gel Capsules of Dr. Reddy's Laboratories Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr. Rama Krishna Bangaru / Assistant Manager, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 02279
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Ibuprofen
MeSH Terms: interventions — Ibuprofen; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental): Ibuprofen 200 mg gel Capsules of Dr. Reddy's laboratories Limited
  Interventions: Drug: Ibuprofen
- Advil (Active Comparator): Advil liquigels 200 mg gel capsules of Wyeth Consumer Healthcare
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 200 mg gel capsules of Dr. Reddy's Laboratories Limited
  Other Names: Advil liquigels 200 mg gel capsules

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of ibuprofen 200 mg gelcaps (test) versus Advil liquigels (reference) administered as 1 x 200 mg gelcap under fasting conditions.

DETAILED DESCRIPTION:
Randomized, 2-way crossover, bioequivalence study of Ibuprofen 200 mg gel capsules and Advil liquigels 200 mg gel caps administered as 1 x 200 mg gel capsule in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be females and/or males, smokers and/or non-smokers, 18 years of age and older.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV) at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90 mmHg; or heart rate less than 50 or over 100 bpm) at screening.
* Subjects with Body Mass Index (BMI) ≥30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* History of allergic reactions to ibuprofen or other nonsteroidal anti- inflammatory drug NSAIDs (e.g. aspirin, diclofenac,diflunisal, etodolac, ketoprofen, fenoprofen, floctafenine, flurbiprofen, indomethacin,ketorolac, mefenamic acid, nabumetone, naproxen, oxaprozin, piroxicam, salsalate, sulindac, tenoxicam, tiaprofenic acid and tolmetin).
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin;examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin,ketoconazole, Mono Amine Oxidase (MAO) inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* History or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug.
* Any history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:

  * less than 300 mL of whole blood within 30 days or
  * 300 mL to 500 mL of whole blood within 45 days or
  * more than 500 mL of whole blood within 56 days
* Subjects who have consumed food or beverages containing grapefruit (e.g. fresh, canned,or frozen) within 7 days prior to administration of the study medication.
* Subjects with history or known presence of active peptic ulcer or heartburn.
* Subjects with history or known presence of gastrointestinal bleeding.
* Subjects with history or known presence of bronchospastic reactivity (e.g. asthma).

For females:

* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).
* Female subjects of childbearing potential who have had unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. The acceptable methods of contraception are:

  * Condom + spermicide
  * Diaphragm + spermicide
  * Intrauterine contraceptive device (placed at least 4 weeks prior to study drug administration).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2002-11; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Study Director — Anapharm
Locations (1):
- Anaphann Inc., Québec, Canada